CLINICAL TRIAL: NCT01503268
Title: Atrial Fibrillation After Catheter Versus Thoracoscopic Ablation Using Patient Activated Implantable Loop Recorders
Brief Title: Atrial Fibrillation After Catheter Versus Thoracoscopic Ablation Using Patient Activated Implantable Loop Recorders: The ACTUAL Study
Acronym: ACTUAL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study methodology redesigned
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Principal Investigator, Neil Sulke, Consultant Cardiologist, Eastbourne General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTUAL 1.0
Record Dates: First submitted 2011-12-30; First posted 2012-01-04 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation; Percutaneous ablation; Minimally-invasive thoracoscopic ablation; Implantable loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Percutaneous ablation (Active Comparator)
  Interventions: Device: Implantation of implantable loop recorder; Procedure: Percutaneous ablation of atrial fibrillation
- Surgical ablation (Active Comparator)
  Interventions: Device: Implantation of implantable loop recorder; Procedure: Surgical ablation of atrial fibrillation
- DCCV (Active Comparator): Direct current cardioversion
  Interventions: Device: Implantation of implantable loop recorder

INTERVENTIONS:
Device: Implantation of implantable loop recorder — An implantable loop recorder (ILR) will be used to assess atrial fibrillation(AF) before and after DCCV or ablation, unless there is a pre-existing ILR or permanent pacemaker capable of continuous monitoring for occurrence of AF.
Procedure: Percutaneous ablation of atrial fibrillation — Catheter-based percutaneous ablation of atrial fibrillation
  Arms: Percutaneous ablation
Procedure: Surgical ablation of atrial fibrillation — Minimally-invasive thoracoscopic surgical ablation of atrial fibrillation
  Arms: Surgical ablation

SUMMARY:
Atrial fibrillation (AF) is a common but often distressing condition. It can be treated with medications, but these are not always effective or tolerated. Ablation is a well-recognised technique that is recommended for those with symptomatic AF who have failed medical therapy.

Ablation can be performed in a number of ways. In percutaneous ablation, ablation is performed via tiny punctures in the skin in the groin. In minimally-invasive thoracoscopic ablation, ablation is performed under general anaesthetic via very small incisions in the chest wall.

Because AF can be intermittent, the only reliable way to look for it is with long-term ECG monitoring. A safe and practical way to do this is to use implantable loop recorders (ILRs).

In this study, the investigators are trying to see if minimally-invasive thoracoscopic ablation is better than percutaneous ablation, and in turn if they are better than Direct current cardioversion (DCCV), using ILRs to monitor AF.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic persistent atrial fibrillation
* Age over 18 years
* Informed consent

Exclusion Criteria:

* Pre-existing ILRs or permanent pacemakers that do not allow for continuous monitoring for AF occurrence, or are not MRI safe.
* Patients unable to undergo general anaesthesia for AF ablation.
* Previous cardiac surgery, such as coronary artery bypass grafting or valvular surgery
* Previous thoracic surgery
* Participation in a conflicting study
* Participants who are mentally incapacitated and cannot consent or comply with follow-up
* Pregnancy
* Other cardiac rhythm disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in AF burden after ablation | One year
  Reduction in proportion of time in atrial fibrillation as detected by an implantable loop recorder
Time to recurrence of persistent AF | 1 year

SECONDARY OUTCOMES:
Time to recurrence of atrial fibrillation after ablation | One year
  Time to first detected episode of atrial fibrillation after ablation, outside a 3 month blanking period
Time to recurrence of symptomatic atrial fibrillation after ablation | One year
  Time to first detected symptomatic episode of atrial fibrillation after ablation, outside a 3 month blanking period
New MRI-detected subclinical cerebral ischaemia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: A N Sulke, MD, Principal Investigator — Eastbourne General Hospital; S S Furniss, MD, Principal Investigator — Eastbourne General Hospital
Locations (2):
- United Kingdom (2):
  - Royal Sussex County Hospital, Brighton, East Sussex
  - Eastbourne District General Hospital, Eastbourne, East Sussex